CLINICAL TRIAL: NCT00081328
Title: Studies to Treat Or Prevent Pediatric Type 2 Diabetes (STOPP-T2D) Treatment Options for Type 2 Diabetes in Adolescents and Youth (TODAY) Clinical Trial
Brief Title: Treatment Options for Type 2 Diabetes in Adolescents and Youth (TODAY)
Acronym: TODAY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IND - DK61230-TODAY; U01DK061230 (NIH)
Record Dates: First submitted 2004-04-08; First posted 2004-04-12 (Estimated); Results first posted 2014-12-16 (Estimated); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Metformin alone
  Interventions: Drug: Metformin
- 2 (Experimental): Metformin + Rosiglitazone
  Interventions: Drug: Metformin; Drug: Rosiglitazone
- 3 (Experimental): Metformin + Lifestyle Program
  Interventions: Drug: Metformin; Behavioral: Lifestyle Program

INTERVENTIONS:
Drug: Metformin — capsule, 1000 mg bid
Drug: Rosiglitazone — capsule, 4 mg bid
  Arms: 2
Behavioral: Lifestyle Program — a lifestyle change (LC) phase of weekly sessions for months 1-6, followed by a bi-weekly lifestyle maintenance (LM) phase through months 7-12, and a continued contact (CC) phase from months 13 through the end of the study. The CC phase sessions are scheduled monthly for the initial 12 months (study months 13-24) and then quarterly or 4 times a year to the end of the study
  Arms: 3

SUMMARY:
The National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) of the National Institutes of Health (NIH) has sponsored a consortium of investigators to conduct a clinical treatment trial, Treatment Options for type 2 Diabetes in Adolescents and Youth (TODAY).

The primary objective of the TODAY trial is to compare the efficacy of three treatment arms on time to treatment failure based on glycemic control. The secondary aims are to:

* compare and evaluate the safety of the three treatment arms;
* compare the effects of the three treatments on the pathophysiology of type 2 diabetes (T2D) with regards to beta cell function and insulin resistance, body composition, nutrition, physical activity and aerobic fitness, cardiovascular risk factors, microvascular complications, quality of life, and psychological outcomes;
* evaluate the influence of individual and family behaviors on treatment response; and
* compare the relative cost effectiveness of the three treatment arms.

The three treatment regimens are: (1) metformin alone, (2) metformin plus rosiglitazone, and (3) metformin plus an intensive lifestyle intervention called the TODAY Lifestyle Program (TLP). The study recruits patients over a three-year period and follows patients for a minimum of two years. Patients are randomized within two years of the diagnosis of T2D.

DETAILED DESCRIPTION:
T2DM has dramatically increased throughout the world in many ethnic groups and among people with diverse social and economic backgrounds. Over the last decade, the increase in the number of children and youth with T2DM has been labeled an "epidemic". Before the 1990s, it was rare for most pediatric centers to have patients with T2DM. By 1994, T2DM patients represented up to 16% of new cases of diabetes in children in urban areas, and by 1999, depending on geographic location, the range of percent of new cases due to T2DM was between 8-45% and disproportionately represented in minority populations.

T2DM in children and youth, as in adults, is due to the combination of insulin resistance and relative β-cell failure. It appears that there are a host of genetic and environmental risk factors for insulin resistance and limited β-cell reserve. The epidemic of pediatric T2DM is coincident with the rise in the number of children who are overweight or at risk for overweight and with a decrease in the physical activity pattern of youth. There has been a strong association between T2DM and the onset of puberty, a positive family history of T2DM, and elements of the metabolic syndrome such as acanthosis nigricans and polycystic ovarian syndrome (PCOS).

Preceding the development of frank diabetes, children and youth experience a period of prediabetes. Prediabetes is defined as either elevated fasting glucose or impaired glucose tolerance. Despite the dramatic increase in the number of cases of prediabetes and T2DM in pediatric populations, there have been no published large-scale studies investigating the pathophysiology, treatment, and complications of these disorders in children and youth. The long-term complications and costs associated with T2DM make such studies imperative. Between 1997 and 2002, the estimated cost of diabetes with regard to direct medical cost increased from $44 billion to $92 billion, and the total cost increased from $98 billion to $132 billion. The vast majority of monies are spent on the long-term complications of this disorder. Since the long-term microvascular and cardiovascular complications relate to duration of diabetes and to control of glycemia, it could be hypothesized that the increasing number of children and youth diagnosed with T2DM, if not effectively treated, could dramatically add to the economic burden of this disease over the ensuing decades.

Except in American Indian youth, there are no population-based data available with regard to prevalence of T2DM. Instead, only clinic-based reports indicate that there has been a tremendous increase in the number of children and adolescents with T2DM. T2DM occurs almost exclusively in children and youth who are overweight or at risk for overweight (BMI > 85th percentile for age). At the time of diagnosis, most pediatric patients are in the midst of Tanner Stage 2-4 puberty. Puberty contributes to insulin resistance due to augmentation of growth hormone secretion, and if these normal pubertal physiologic changes are not compensated for by increased insulin secretion, frank diabetes will develop. Half to three-quarters of patients have a parent and close to ninety percent have at least one first or second degree relative with T2DM. The clinical presentation of T2DM in youth ranges from mild asymptomatic hyperglycemia to severe ketoacidosis. In those who present with clinical symptoms due to hyperglycemia, glycosuria and weight loss are present in 20-40%, ketonuria is present in 33% and ketoacidosis is found in 5-10%. Patients without clinical symptoms are diagnosed as the result of routine blood or urine testing during a health care visit or by investigating a variety of complaints such as chronic infection, sleep apnea, hyperlipidemia, hypertension, and hirsutism or irregular periods associated with PCOS. It may be difficult to distinguish T1DM from T2DM at presentation. The absence of autoantibodies is a prerequisite for the diagnosis of T2DM. In addition, evidence of residual insulin secretion is suggestive of T2DM rather than T1DM.

Patients with T2DM have dual abnormalities of insulin resistance and insulin deficiency. It is hypothesized that to achieve the level of glycemic control required to optimize long-term outcome and decrease or prevent microvascular complications, treatment regimens should theoretically be designed to improve insulin resistance and preserve residual β-cell function. The available anti-diabetic agents have not been adequately evaluated in pediatric patients. This is particularly relevant with regard to using combination therapy to improve glycemic control or lifestyle interventions aimed at obesity and sedentary behavior.

ELIGIBILITY:
Inclusion Criteria (during Screening and Run-in period):

* Diabetes by ADA criteria (laboratory determinations of fasting glucose ≥ 126 mg/dL, random glucose ≥ 200 mg/dL, or two-hour OGTT glucose ≥ 200 mg/dL) documented and confirmed in medical record. For patients diagnosed with diabetes during screening who have a normal fasting glucose but an elevated two-hour glucose during an OGTT, the HbA1c must be ≥ 6%.
* Duration since diagnosis less than two years by date of randomization.
* BMI ≥ 85th percentile documented at time of diagnosis or at screening.
* Fasting C-peptide at screening (drawn at least one week after treatment for ketosis or acidosis, if applicable) > 0.6 ng/mL.
* Absence of pancreatic autoimmunity (both GAD and ICA512 negative).
* Age 10-17, with randomization prior to 18th birthday.
* Signed informed consent/assent forms for the pre-randomization period.
* A family member or adult closely involved in the daily activities of the child agrees to participate in the child's treatment.
* Fluency in English or Spanish for both child and family member.
* Patient and family able to fully participate in trial protocol in the opinion of the investigator.

Exclusion Criteria (during Screening and Run-in period):

* Participating in another interventional research study protocol in the past 30 days.
* Genetic syndrome or disorder known to affect glucose tolerance other than diabetes.
* Patient on inhaled steroids at dose above 1000 mcg daily Flovent equivalent.
* Patient on a course of oral steroids within the last 60 days or on oral steroids more than 20 days during the past year.
* Patient on medication(s) that are known to affect insulin sensitivity or secretion within the last 30 days.
* Patient on medication(s) that are known to cause weight gain within the last 30 days.
* Patient on any weight-loss medication(s) within the last 30 days.
* Patient on medication(s) known to affect the metabolism of study drug.
* Inability to comprehend the lowest grade level at which lifestyle intervention materials are prepared, for both child and participating family member.
* Females who are pregnant, planning to become pregnant within two years of enrollment, or who admit sexual activity without appropriate contraception.
* Calculated creatinine clearance < 70 mL/min.
* Any transaminase > 2.5 ULN. If any transaminase 1.5-2.5 times ULN, then patient must be appropriately evaluated by PCP (minimum evaluation includes ceruloplasmin level, alpha-1 antitrypsin phenotype, ANA, anti-smooth muscle antibody, anti-LKM antibody, anti-HCV, and anti-HBc total antibody not IgM, iron, and TIBC) and is eligible if all other causes for elevation are ruled out and it is presumed due only to non-alcoholic fatty liver disease (NAFLD).
* Diabetic ketoacidosis (DKA) at any time after diagnosis unless only a single episode of DKA related to a significant medical illness.
* Physical limitations preventing patient from being randomized to the lifestyle intervention.
* Patient plans to leave the geographic area within one calendar year.
* Abnormal reticulocyte count or HbA1c chromatogram at time of screening.
* Admitted use of anabolic steroids within the past 60 days.
* Other significant organ system illness or condition (including psychiatric or developmental disorder) that would prevent participation in the opinion of the investigator.
* Patient participates in a formal weight-loss program.

Inclusion Criteria (post Run-in and Randomization):

* Duration since diagnosis less than 2 years at randomization.
* HbA1c < 8% on metformin alone.
* Age 10-17, with randomization before patient is 18 years old.
* Signed consent/assent forms for randomization and the post-randomization phase.
* A family member or adult closely involved in the daily activities of the child agrees to participate in the child's treatment.
* Fluency in English or Spanish for both child and family member.
* Patient and family able to fully participate in trial protocol in the opinion of the investigator.

Exclusion Criteria (post Run-in and Randomization):

* Refractory hypertension: average systolic blood pressure ≥ 150 mmHg or average diastolic blood pressure ≥ 95 mmHg despite appropriate medical therapy.
* Refractory hyperlipidemia: total cholesterol > 300 mg/dL or LDL > 190 mg/dL or triglycerides > 800 mg/dL, despite appropriate medical therapy.
* Refractory anemia: hematocrit < 30% or hemoglobin < 10 gm/dL despite appropriate medical therapy.
* Patient on a thiazolidinedione (TZD) within the last 12 weeks.
* Patient on non-study diabetes medications within the past 6 weeks.
* Patient on inhaled steroids at dose above 1000 mcg daily Flovent equivalent.
* Patient on a course of oral steroids within the last 60 days or on oral steroids more than 20 days during the past year.
* Patient on medication(s) that are known to affect insulin sensitivity or secretion within the last 30 days.
* Patient on medication(s) that are known to cause weight gain within the last 30 days.
* Patient on any weight-loss medication(s) within the last 30 days.
* Patient on medication(s) known to affect the metabolism of study drug.
* Inability to comprehend the lowest grade level at which lifestyle intervention materials are prepared, for both child and participating family member, assessed by mastery of standard diabetes education program administered during run-in.
* Inability to comply with requirements of study during run-in period.
* Females who are pregnant, planning to become pregnant within two years of enrollment, or who admit sexual activity without appropriate contraception.
* Calculated creatinine clearance < 70 mL/min.
* Physical limitations preventing patient from being randomized to the lifestyle intervention.
* Patient plans to leave the geographic area within one calendar year.
* Admitted use of anabolic steroids within 60 days.
* Other significant organ system illness or condition (including psychiatric or developmental disorder) that would prevent participation in the opinion of the investigator.
* Patient participates in a formal weight loss program.
* Episode of DKA during the run-in.30.
* Edema at the time of randomization (a participant who experiences edema during run-in must have recovered within 2 weeks and be edema free for 1 week prior to randomization).

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 699 (Actual)
Dates: Start 2004-05; Primary Completion 2011-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phil Zeitler, MD, PhD, Principal Investigator — University of Colorado, Denver; Kathryn Hirst, PhD, Principal Investigator — George Washington University
Locations (16):
- United States (16):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of Colorado Health Sciences Center, The Children's Hospital, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - George Washington University Biostatistics Center, Rockville, Maryland
  - Massachusetts General Hospital Diabetes Center, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Saint Louis University Health Sciences Center, St Louis, Missouri
  - Washington University Department of Pediatrics, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Case Western Reserve, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository
URL: https://repository.niddk.nih.gov/studies/today/?query=today

REFERENCES:
- [Background] TODAY Study Group; Zeitler P, Epstein L, Grey M, Hirst K, Kaufman F, Tamborlane W, Wilfley D. Treatment options for type 2 diabetes in adolescents and youth: a study of the comparative efficacy of metformin alone or in combination with rosiglitazone or lifestyle intervention in adolescents with type 2 diabetes. Pediatr Diabetes. 2007 Apr;8(2):74-87. doi: 10.1111/j.1399-5448.2007.00237.x. PMID 17448130
- [Background] Songer T, Glazner J, Coombs LP, Cuttler L, Daniel M, Estrada S, Klingensmith G, Kriska A, Laffel L, Zhang P; the TODAY Study Group. Examining the economic costs related to lifestyle and pharmacological interventions in youth with Type 2 diabetes. Expert Rev Pharmacoecon Outcomes Res. 2006 Jun 1;6(3):315-324. doi: 10.1586/14737167.6.3.315. PMID 19774104
- [Background] Grey M, Schreiner B, Pyle L. Development of a diabetes education program for youth with type 2 diabetes. Diabetes Educ. 2009 Jan-Feb;35(1):108-16. doi: 10.1177/0145721708325156. PMID 19244566
- [Background] TODAY Study Group. Design of a family-based lifestyle intervention for youth with type 2 diabetes: the TODAY study. Int J Obes (Lond). 2010 Feb;34(2):217-26. doi: 10.1038/ijo.2009.195. Epub 2009 Oct 13. PMID 19823189
- [Background] Larkin ME, McGuigan P, Richards D, Blumenthal K, Milaszewski K, Higgins L, Schanuel J, Long C. Collaborative Staffing Model for Multiple Sites: Reducing the challenges of study coordination in complex, multi-site clinical trials. Appl Clin Trials. 2011 Jan 1;20(1):30-35. PMID 24955003
- [Background] Chadwick JQ, Copeland KC, Daniel MR, Erb-Alvarez JA, Felton BA, Khan SI, Saunkeah BR, Wharton DF, Payan ML. Partnering in research: a national research trial exemplifying effective collaboration with American Indian Nations and the Indian Health Service. Am J Epidemiol. 2014 Dec 15;180(12):1202-7. doi: 10.1093/aje/kwu246. Epub 2014 Nov 11. PMID 25389367
- [Background] Chadwick JQ, Van Buren DJ, Morales E, Timpson A, Abrams EL, Syme A, Preske J, Mireles G, Anderson B, Grover N, Laffel L. Structure to utilize interventionists' implementation experiences of a family-based behavioral weight management program to enhance the dissemination of the standardized intervention: The TODAY study. Clin Trials. 2017 Aug;14(4):406-412. doi: 10.1177/1740774517707727. Epub 2017 May 9. PMID 28486851
- [Background] Chadwick JQ, Copeland KC, Branam DE, Erb-Alvarez JA, Khan SI, Peercy MT, Rogers ME, Saunkeah BR, Tryggestad JB, Wharton DF. Genomic Research and American Indian Tribal Communities in Oklahoma: Learning From Past Research Misconduct and Building Future Trusting Partnerships. Am J Epidemiol. 2019 Jul 1;188(7):1206-1212. doi: 10.1093/aje/kwz062. PMID 31081852
- [Background] Songer TJ, Haymond MW, Glazner JE, Klingensmith GJ, Laffel LM, Zhang P, Hirst K; TODAY Study Group. Healthcare and associated costs related to type 2 diabetes in youth and adolescence: the TODAY clinical trial experience. Pediatr Diabetes. 2019 Sep;20(6):702-711. doi: 10.1111/pedi.12869. Epub 2019 Jun 6. PMID 31119838
- [Result] Klingensmith GJ, Pyle L, Arslanian S, Copeland KC, Cuttler L, Kaufman F, Laffel L, Marcovina S, Tollefsen SE, Weinstock RS, Linder B; TODAY Study Group. The presence of GAD and IA-2 antibodies in youth with a type 2 diabetes phenotype: results from the TODAY study. Diabetes Care. 2010 Sep;33(9):1970-5. doi: 10.2337/dc10-0373. Epub 2010 Jun 2. PMID 20519658
- [Result] Copeland KC, Zeitler P, Geffner M, Guandalini C, Higgins J, Hirst K, Kaufman FR, Linder B, Marcovina S, McGuigan P, Pyle L, Tamborlane W, Willi S; TODAY Study Group. Characteristics of adolescents and youth with recent-onset type 2 diabetes: the TODAY cohort at baseline. J Clin Endocrinol Metab. 2011 Jan;96(1):159-67. doi: 10.1210/jc.2010-1642. Epub 2010 Oct 20. PMID 20962021
- [Result] TODAY Study Group; Wilfley D, Berkowitz R, Goebel-Fabbri A, Hirst K, Ievers-Landis C, Lipman TH, Marcus M, Ng D, Pham T, Saletsky R, Schanuel J, Van Buren D. Binge eating, mood, and quality of life in youth with type 2 diabetes: baseline data from the today study. Diabetes Care. 2011 Apr;34(4):858-60. doi: 10.2337/dc10-1704. Epub 2011 Feb 28. PMID 21357794
- [Result] Anderson BJ, Edelstein S, Abramson NW, Katz LE, Yasuda PM, Lavietes SJ, Trief PM, Tollefsen SE, McKay SV, Kringas P, Casey TL, Marcus MD. Depressive symptoms and quality of life in adolescents with type 2 diabetes: baseline data from the TODAY study. Diabetes Care. 2011 Oct;34(10):2205-7. doi: 10.2337/dc11-0431. Epub 2011 Aug 11. PMID 21836107
- [Result] Laffel L, Chang N, Grey M, Hale D, Higgins L, Hirst K, Izquierdo R, Larkin M, Macha C, Pham T, Wauters A, Weinstock RS; TODAY Study Group. Metformin monotherapy in youth with recent onset type 2 diabetes: experience from the prerandomization run-in phase of the TODAY study. Pediatr Diabetes. 2012 Aug;13(5):369-75. doi: 10.1111/j.1399-5448.2011.00846.x. Epub 2012 Feb 27. PMID 22369102
- [Result] Bacha F, Pyle L, Nadeau K, Cuttler L, Goland R, Haymond M, Levitsky L, Lynch J, Weinstock RS, White NH, Caprio S, Arslanian S; TODAY Study Group. Determinants of glycemic control in youth with type 2 diabetes at randomization in the TODAY study. Pediatr Diabetes. 2012 Aug;13(5):376-83. doi: 10.1111/j.1399-5448.2011.00841.x. Epub 2012 Feb 15. PMID 22332798
- [Result] TODAY Study Group; Zeitler P, Hirst K, Pyle L, Linder B, Copeland K, Arslanian S, Cuttler L, Nathan DM, Tollefsen S, Wilfley D, Kaufman F. A clinical trial to maintain glycemic control in youth with type 2 diabetes. N Engl J Med. 2012 Jun 14;366(24):2247-56. doi: 10.1056/NEJMoa1109333. Epub 2012 Apr 29. PMID 22540912
- [Result] Kriska A, Delahanty L, Edelstein S, Amodei N, Chadwick J, Copeland K, Galvin B, El ghormli L, Haymond M, Kelsey M, Lassiter C, Mayer-Davis E, Milaszewski K, Syme A. Sedentary behavior and physical activity in youth with recent onset of type 2 diabetes. Pediatrics. 2013 Mar;131(3):e850-6. doi: 10.1542/peds.2012-0620. Epub 2013 Feb 11. PMID 23400602
- [Result] Delahanty L, Kriska A, Edelstein S, Amodei N, Chadwick J, Copeland K, Galvin B, El Ghormli L, Haymond M, Kelsey MM, Lassiter C, Milaszewski K, Syme A, Mayer-Davis E. Self-reported dietary intake of youth with recent onset of type 2 diabetes: results from the TODAY study. J Acad Nutr Diet. 2013 Mar;113(3):431-439. doi: 10.1016/j.jand.2012.11.015. PMID 23438494
- [Result] TODAY Study Group. Rapid rise in hypertension and nephropathy in youth with type 2 diabetes: the TODAY clinical trial. Diabetes Care. 2013 Jun;36(6):1735-41. doi: 10.2337/dc12-2420. PMID 23704672
- [Result] TODAY Study Group. Treatment effects on measures of body composition in the TODAY clinical trial. Diabetes Care. 2013 Jun;36(6):1742-8. doi: 10.2337/dc12-2534. PMID 23704673
- [Result] TODAY Study Group. Effects of metformin, metformin plus rosiglitazone, and metformin plus lifestyle on insulin sensitivity and beta-cell function in TODAY. Diabetes Care. 2013 Jun;36(6):1749-57. doi: 10.2337/dc12-2393. PMID 23704674
- [Result] TODAY Study Group. Lipid and inflammatory cardiovascular risk worsens over 3 years in youth with type 2 diabetes: the TODAY clinical trial. Diabetes Care. 2013 Jun;36(6):1758-64. doi: 10.2337/dc12-2388. PMID 23704675
- [Result] TODAY Study Group. Safety and tolerability of the treatment of youth-onset type 2 diabetes: the TODAY experience. Diabetes Care. 2013 Jun;36(6):1765-71. doi: 10.2337/dc12-2390. PMID 23704676
- [Result] TODAY Study Group. Retinopathy in youth with type 2 diabetes participating in the TODAY clinical trial. Diabetes Care. 2013 Jun;36(6):1772-4. doi: 10.2337/dc12-2387. PMID 23704677
- [Result] Levitt Katz L, Gidding SS, Bacha F, Hirst K, McKay S, Pyle L, Lima JA; TODAY Study Group. Alterations in left ventricular, left atrial, and right ventricular structure and function to cardiovascular risk factors in adolescents with type 2 diabetes participating in the TODAY clinical trial. Pediatr Diabetes. 2015 Feb;16(1):39-47. doi: 10.1111/pedi.12119. Epub 2014 Jan 22. PMID 24450390
- [Result] Narasimhan S, Weinstock RS. Youth-onset type 2 diabetes mellitus: lessons learned from the TODAY study. Mayo Clin Proc. 2014 Jun;89(6):806-16. doi: 10.1016/j.mayocp.2014.01.009. Epub 2014 Apr 3. PMID 24702733
- [Result] Walders-Abramson N, Venditti EM, Ievers-Landis CE, Anderson B, El Ghormli L, Geffner M, Kaplan J, Koontz MB, Saletsky R, Payan M, Yasuda P; Treatment Options for Type 2 Diabetes in Adolescents and Youth (TODAY) Study Group. Relationships among stressful life events and physiological markers, treatment adherence, and psychosocial functioning among youth with type 2 diabetes. J Pediatr. 2014 Sep;165(3):504-508.e1. doi: 10.1016/j.jpeds.2014.05.020. Epub 2014 Jun 16. PMID 24948348
- [Result] Tryggestad JB, Willi SM. Complications and comorbidities of T2DM in adolescents: findings from the TODAY clinical trial. J Diabetes Complications. 2015 Mar;29(2):307-12. doi: 10.1016/j.jdiacomp.2014.10.009. Epub 2014 Oct 29. PMID 25468310
- [Result] Weinstock RS, Trief PM, El Ghormli L, Goland R, McKay S, Milaszewski K, Preske J, Willi S, Yasuda PM. Parental Characteristics Associated With Outcomes in Youth With Type 2 Diabetes: Results From the TODAY Clinical Trial. Diabetes Care. 2015 May;38(5):784-92. doi: 10.2337/dc14-2393. Epub 2015 Mar 17. PMID 25784663
- [Result] Weinstock RS, Drews KL, Caprio S, Leibel NI, McKay SV, Zeitler PS; TODAY Study Group. Metabolic syndrome is common and persistent in youth-onset type 2 diabetes: Results from the TODAY clinical trial. Obesity (Silver Spring). 2015 Jul;23(7):1357-61. doi: 10.1002/oby.21120. Epub 2015 Jun 5. PMID 26047470
- [Result] Ievers-Landis CE, Walders-Abramson N, Amodei N, Drews KL, Kaplan J, Levitt Katz LE, Lavietes S, Saletsky R, Seidman D, Yasuda P; Treatment Options for Type 2 Diabetes in Adolescents and Youth (TODAY) Study Group. Longitudinal Correlates of Health Risk Behaviors in Children and Adolescents with Type 2 Diabetes. J Pediatr. 2015 May;166(5):1258-1264.e3. doi: 10.1016/j.jpeds.2015.01.019. Epub 2015 Feb 20. PMID 25702853
- [Result] Larkin ME, Walders-Abramson N, Hirst K, Keady J, Ievers-Landis CE, Venditti EM, Yasuda PM. Effects of comorbid conditions on health-related quality of life in youth with Type 2 diabetes: the TODAY clinical trial. Diabetes Manag (Lond). 2015 Nov;5(6):431-439. doi: 10.2217/dmt.15.35. PMID 27057209
- [Result] Zeitler P, Hirst K, Copeland KC, El Ghormli L, Levitt Katz L, Levitsky LL, Linder B, McGuigan P, White NH, Wilfley D; TODAY Study Group. HbA1c After a Short Period of Monotherapy With Metformin Identifies Durable Glycemic Control Among Adolescents With Type 2 Diabetes. Diabetes Care. 2015 Dec;38(12):2285-92. doi: 10.2337/dc15-0848. Epub 2015 Nov 4. PMID 26537182
- [Result] Walders-Abramson N, Anderson B, Larkin ME, Chang N, Venditti E, Bzdick S, Tryggestad JB, Tan K, Geffner ME, Hirst K. Benefits and barriers to participating in longitudinal research of youth-onset type 2 diabetes: Results from the TODAY retention survey. Clin Trials. 2016 Apr;13(2):240-3. doi: 10.1177/1740774515613949. Epub 2015 Nov 3. PMID 26531295
- [Result] Chernausek SD, Arslanian S, Caprio S, Copeland KC, El ghormli L, Kelsey MM, Koontz MB, Orsi CM, Wilfley D. Relationship Between Parental Diabetes and Presentation of Metabolic and Glycemic Function in Youth With Type 2 Diabetes: Baseline Findings From the TODAY Trial. Diabetes Care. 2016 Jan;39(1):110-7. doi: 10.2337/dc15-1557. Epub 2015 Nov 17. PMID 26577415
- [Result] Klingensmith GJ, Pyle L, Nadeau KJ, Barbour LA, Goland RS, Willi SM, Linder B, White NH; TODAY Study Group. Pregnancy Outcomes in Youth With Type 2 Diabetes: The TODAY Study Experience. Diabetes Care. 2016 Jan;39(1):122-9. doi: 10.2337/dc15-1206. Epub 2015 Dec 1. PMID 26628417
- [Result] Kelsey MM, Geffner ME, Guandalini C, Pyle L, Tamborlane WV, Zeitler PS, White NH; Treatment Options for Type 2 Diabetes in Adolescents and Youth Study Group. Presentation and effectiveness of early treatment of type 2 diabetes in youth: lessons from the TODAY study. Pediatr Diabetes. 2016 May;17(3):212-21. doi: 10.1111/pedi.12264. Epub 2015 Feb 17. PMID 25690268
- [Result] Rockette-Wagner B, Storti KL, Edelstein S, Delahanty LM, Galvin B, Jackson A, Kriska AM. Measuring Physical Activity and Sedentary Behavior in Youth with Type 2 Diabetes. Child Obes. 2017 Feb;13(1):72-77. doi: 10.1089/chi.2015.0151. Epub 2016 Feb 9. PMID 26859798
- [Result] Arslanian S, El Ghormli L, Bacha F, Caprio S, Goland R, Haymond MW, Levitsky L, Nadeau KJ, White NH, Willi SM; TODAY Study Group. Adiponectin, Insulin Sensitivity, beta-Cell Function, and Racial/Ethnic Disparity in Treatment Failure Rates in TODAY. Diabetes Care. 2017 Jan;40(1):85-93. doi: 10.2337/dc16-0455. Epub 2016 Nov 1. PMID 27803118
- [Result] Marcus MD, Wilfley DE, El Ghormli L, Zeitler P, Linder B, Hirst K, Ievers-Landis CE, van Buren DJ, Walders-Abramson N; TODAY Study Group. Weight change in the management of youth-onset type 2 diabetes: the TODAY clinical trial experience. Pediatr Obes. 2017 Aug;12(4):337-345. doi: 10.1111/ijpo.12148. Epub 2016 May 10. PMID 27161901
- [Result] Gandica R, Zeitler P. Update on Youth-Onset Type 2 Diabetes: Lessons Learned from the Treatment Options for Type 2 Diabetes in Adolescents and Youth Clinical Trial. Adv Pediatr. 2016 Aug;63(1):195-209. doi: 10.1016/j.yapd.2016.04.013. Epub 2016 Jun 3. No abstract available. PMID 27426901
- [Result] Katz LL, Anderson BJ, McKay SV, Izquierdo R, Casey TL, Higgins LA, Wauters A, Hirst K, Nadeau KJ; TODAY Study Group. Correlates of Medication Adherence in the TODAY Cohort of Youth With Type 2 Diabetes. Diabetes Care. 2016 Nov;39(11):1956-1962. doi: 10.2337/dc15-2296. Epub 2016 Jun 28. PMID 27352955
- [Result] Bacha F, Gidding SS, Pyle L, Levitt Katz L, Kriska A, Nadeau KJ, Lima JAC; Treatment Options for Type 2 Diabetes in Adolescents and Youth (TODAY) Study Group. Relationship of Cardiac Structure and Function to Cardiorespiratory Fitness and Lean Body Mass in Adolescents and Young Adults with Type 2 Diabetes. J Pediatr. 2016 Oct;177:159-166.e1. doi: 10.1016/j.jpeds.2016.06.048. Epub 2016 Aug 4. PMID 27499218
- [Result] Kriska A, El Ghormli L, Copeland KC, Higgins J, Ievers-Landis CE, Levitt Katz LE, Trief PM, Wauters AD, Yasuda PM, Delahanty LM; TODAY Study Group. Impact of lifestyle behavior change on glycemic control in youth with type 2 diabetes. Pediatr Diabetes. 2018 Feb;19(1):36-44. doi: 10.1111/pedi.12526. Epub 2017 Apr 4. PMID 28378429
- [Result] Berkowitz RI, Marcus MD, Anderson BJ, Delahanty L, Grover N, Kriska A, Laffel L, Syme A, Venditti E, Van Buren DJ, Wilfley DE, Yasuda P, Hirst K; TODAY Study Group. Adherence to a lifestyle program for youth with type 2 diabetes and its association with treatment outcome in the TODAY clinical trial. Pediatr Diabetes. 2018 Mar;19(2):191-198. doi: 10.1111/pedi.12555. Epub 2017 Jun 30. PMID 28664624
- [Result] Bjornstad P, Nehus E, El Ghormli L, Bacha F, Libman IM, McKay S, Willi SM, Laffel L, Arslanian S, Nadeau KJ; TODAY Study Group. Insulin Sensitivity and Diabetic Kidney Disease in Children and Adolescents With Type 2 Diabetes: An Observational Analysis of Data From the TODAY Clinical Trial. Am J Kidney Dis. 2018 Jan;71(1):65-74. doi: 10.1053/j.ajkd.2017.07.015. Epub 2017 Nov 20. PMID 29157731
- [Result] Gidding SS, Bacha F, Bjornstad P, Levitt Katz LE, Levitsky LL, Lynch J, Tryggestad JB, Weinstock RS, El Ghormli L, Lima JAC; TODAY Study Group. Cardiac Biomarkers in Youth with Type 2 Diabetes Mellitus: Results from the TODAY Study. J Pediatr. 2018 Jan;192:86-92.e5. doi: 10.1016/j.jpeds.2017.09.012. PMID 29246363
- [Result] Kleinberger JW, Copeland KC, Gandica RG, Haymond MW, Levitsky LL, Linder B, Shuldiner AR, Tollefsen S, White NH, Pollin TI. Monogenic diabetes in overweight and obese youth diagnosed with type 2 diabetes: the TODAY clinical trial. Genet Med. 2018 Jun;20(6):583-590. doi: 10.1038/gim.2017.150. Epub 2017 Oct 12. PMID 29758564
- [Result] Van Buren DJ, Wilfley DE, Marcus MD, Anderson B, Abramson NW, Berkowitz R, Ievers-Landis C, Trief P, Yasuda P, Hirst K; TODAY Study Group. Depressive symptoms and glycemic control in youth with type 2 diabetes participating in the TODAY clinical trial. Diabetes Res Clin Pract. 2018 Jan;135:85-87. doi: 10.1016/j.diabres.2017.11.008. Epub 2017 Nov 13. PMID 29146120
- [Result] Levitt Katz LE, Bacha F, Gidding SS, Weinstock RS, El Ghormli L, Libman I, Nadeau KJ, Porter K, Marcovina S; TODAY Study Group. Lipid Profiles, Inflammatory Markers, and Insulin Therapy in Youth with Type 2 Diabetes. J Pediatr. 2018 May;196:208-216.e2. doi: 10.1016/j.jpeds.2017.12.052. Epub 2018 Feb 2. PMID 29398050
- [Result] Inge TH, Laffel LM, Jenkins TM, Marcus MD, Leibel NI, Brandt ML, Haymond M, Urbina EM, Dolan LM, Zeitler PS; Teen-Longitudinal Assessment of Bariatric Surgery (Teen-LABS) and Treatment Options of Type 2 Diabetes in Adolescents and Youth (TODAY) Consortia. Comparison of Surgical and Medical Therapy for Type 2 Diabetes in Severely Obese Adolescents. JAMA Pediatr. 2018 May 1;172(5):452-460. doi: 10.1001/jamapediatrics.2017.5763. PMID 29532078
- [Result] Venditti EM, Tan K, Chang N, Laffel L, McGinley G, Miranda N, Tryggestad JB, Walders-Abramson N, Yasuda P, Delahanty L; TODAY Study Group. Barriers and strategies for oral medication adherence among children and adolescents with Type 2 diabetes. Diabetes Res Clin Pract. 2018 May;139:24-31. doi: 10.1016/j.diabres.2018.02.001. Epub 2018 Feb 8. PMID 29427697
- [Result] Kelsey MM, Braffett BH, Geffner ME, Levitsky LL, Caprio S, McKay SV, Shah R, Sprague JE, Arslanian SA; TODAY Study Group. Menstrual Dysfunction in Girls From the Treatment Options for Type 2 Diabetes in Adolescents and Youth (TODAY) Study. J Clin Endocrinol Metab. 2018 Jun 1;103(6):2309-2318. doi: 10.1210/jc.2018-00132. PMID 29697830
- [Result] Shah AS, El Ghormli L, Gidding SS, Bacha F, Nadeau KJ, Levitt Katz LE, Tryggestad JB, Leibel N, Hale DE, Urbina EM. Prevalence of arterial stiffness in adolescents with type 2 diabetes in the TODAY cohort: Relationships to glycemic control and other risk factors. J Diabetes Complications. 2018 Aug;32(8):740-745. doi: 10.1016/j.jdiacomp.2018.05.013. Epub 2018 May 25. PMID 29936086
- [Result] Arslanian S, El Ghormli L, Young Kim J, Bacha F, Chan C, Ismail HM, Levitt Katz LE, Levitsky L, Tryggestad JB, White NH; TODAY Study Group. The Shape of the Glucose Response Curve During an Oral Glucose Tolerance Test: Forerunner of Heightened Glycemic Failure Rates and Accelerated Decline in beta-Cell Function in TODAY. Diabetes Care. 2019 Jan;42(1):164-172. doi: 10.2337/dc18-1122. Epub 2018 Nov 19. PMID 30455329
- [Result] Weinstock RS, Braffett BH, McGuigan P, Larkin ME, Grover NB, Walders-Abramson N, Laffel LM, Chan CL, Chang N, Schwartzman BE, Barajas RA, Celona-Jacobs N, Haymond MW; TODAY Study Group. Self-Monitoring of Blood Glucose in Youth-Onset Type 2 Diabetes: Results From the TODAY Study. Diabetes Care. 2019 May;42(5):903-909. doi: 10.2337/dc18-1854. Epub 2019 Mar 4. PMID 30833375
- [Result] Bjornstad P, Laffel L, Lynch J, El Ghormli L, Weinstock RS, Tollefsen SE, Nadeau KJ; TODAY Study Group. Elevated Serum Uric Acid Is Associated With Greater Risk for Hypertension and Diabetic Kidney Diseases in Obese Adolescents With Type 2 Diabetes: An Observational Analysis From the Treatment Options for Type 2 Diabetes in Adolescents and Youth (TODAY) Study. Diabetes Care. 2019 Jun;42(6):1120-1128. doi: 10.2337/dc18-2147. Epub 2019 Apr 9. PMID 30967435
- [Result] Dhaliwal R, Shepherd JA, El Ghormli L, Copeland KC, Geffner ME, Higgins J, Levitsky LL, Nadeau KJ, Weinstock RS, White NH; TODAY Study Group. Changes in Visceral and Subcutaneous Fat in Youth With Type 2 Diabetes in the TODAY Study. Diabetes Care. 2019 Aug;42(8):1549-1559. doi: 10.2337/dc18-1935. Epub 2019 Jun 5. PMID 31167889
- [Result] Bacha F, El Ghormli L, Arslanian S, Zeitler P, Laffel LM, Levitt Katz LE, Gandica R, Chang NT, Sprague JE, Macleish SA; TODAY Study Group. Predictors of response to insulin therapy in youth with poorly-controlled type 2 diabetes in the TODAY trial. Pediatr Diabetes. 2019 Nov;20(7):871-879. doi: 10.1111/pedi.12906. Epub 2019 Aug 27. PMID 31418516
- [Result] Shah AS, El Ghormli L, Vajravelu ME, Bacha F, Farrell RM, Gidding SS, Levitt Katz LE, Tryggestad JB, White NH, Urbina EM. Heart Rate Variability and Cardiac Autonomic Dysfunction: Prevalence, Risk Factors, and Relationship to Arterial Stiffness in the Treatment Options for Type 2 Diabetes in Adolescents and Youth (TODAY) Study. Diabetes Care. 2019 Nov;42(11):2143-2150. doi: 10.2337/dc19-0993. Epub 2019 Sep 9. PMID 31501226
- [Result] Bjornstad P, Hughan K, Kelsey MM, Shah AS, Lynch J, Nehus E, Mitsnefes M, Jenkins T, Xu P, Xie C, Inge T, Nadeau K. Effect of Surgical Versus Medical Therapy on Diabetic Kidney Disease Over 5 Years in Severely Obese Adolescents With Type 2 Diabetes. Diabetes Care. 2020 Jan;43(1):187-195. doi: 10.2337/dc19-0708. Epub 2019 Nov 4. PMID 31685489
- [Result] Shah R, McKay SV, Levitt Katz LE, El Ghormli L, Anderson BJ, Casey TL, Higgins L, Izquierdo R, Wauters AD, Chang N; TODAY Study Group. Adherence to multiple medications in the TODAY (Treatment Options for type 2 Diabetes in Adolescents and Youth) cohort: effect of additional medications on adherence to primary diabetes medication. J Pediatr Endocrinol Metab. 2020 Feb 25;33(2):191-198. doi: 10.1515/jpem-2019-0315. PMID 31809265
- [Result] Kaar JL, Schmiege SJ, Drews K, Higgins J, Walders-Abramson N, Isganaitis E, Willi SM, Marcus MD, Zeitler PS, Kelsey MM. Evaluation of the longitudinal change in health behavior profiles across treatment groups in the TODAY clinical trial. Pediatr Diabetes. 2020 Mar;21(2):224-232. doi: 10.1111/pedi.12976. Epub 2020 Jan 6. PMID 31886931
- [Result] Arslanian S, El Ghormli L, Haymond MH, Chan CL, Chernausek SD, Gandica RG, Gubitosi-Klug R, Levitsky LL, Siska M, Willi SM; TODAY Study Group. Beta cell function and insulin sensitivity in obese youth with maturity onset diabetes of youth mutations vs type 2 diabetes in TODAY: Longitudinal observations and glycemic failure. Pediatr Diabetes. 2020 Jun;21(4):575-585. doi: 10.1111/pedi.12998. Epub 2020 Mar 3. PMID 32064729
- [Result] Tryggestad JB, Shah RD, Braffett BH, Bacha F, Gidding SS, Gubitosi-Klug RA, Shah AS, Urbina EM, Levitt Katz LE; TODAY Study Group. Circulating adhesion molecules and associations with HbA1c, hypertension, nephropathy, and retinopathy in the Treatment Options for type 2 Diabetes in Adolescent and Youth study. Pediatr Diabetes. 2020 Sep;21(6):923-931. doi: 10.1111/pedi.13062. Epub 2020 Jul 2. PMID 32501612
- [Result] Ryder JR, Xu P, Nadeau KJ, Kelsey MM, Xie C, Jenkins T, Inge TH, Bjornstad P. Effect of surgical versus medical therapy on estimated cardiovascular event risk among adolescents with type 2 diabetes and severe obesity. Surg Obes Relat Dis. 2021 Jan;17(1):23-33. doi: 10.1016/j.soard.2020.09.002. Epub 2020 Sep 9. PMID 33071178
- [Derived] Levitt Katz LE, El Ghormli LK, Nadeau KJ, Shah A, Higgins J, Kutney K, Gubitosi-Klug R, Burke B, Mokhlesi B; TODAY Study Group. Obstructive sleep apnea, glycemic control, and cardiovascular risk in young adults with youth-onset type 2 diabetes: results from the TODAY study. J Clin Sleep Med. 2025 Nov 1;21(11):1925-1933. doi: 10.5664/jcsm.11784. PMID 40566988
- [Derived] Nadeau KJ, Arslanian SA, Bacha F, Caprio S, Chao LC, Farrell R, Hughan KS, Rayas M, Tung M, Cross K, El Ghormli L; TODAY Study Group. Insulin clearance at randomisation and in response to treatment in youth with type 2 diabetes: a secondary analysis of the TODAY randomised clinical trial. Diabetologia. 2025 Mar;68(3):676-687. doi: 10.1007/s00125-024-06327-w. Epub 2024 Dec 20. PMID 39706874
- [Derived] Pyle L, Choi YJ, Narongkiatikhun P, Sharma K, Waikar S, Layton A, Tommerdahl KL, de Boer I, Vigers T, Nelson RG, Lynch J, Brosius F 3rd, Saulnier PJ, Goodrich JA, Tryggestad JB, Isganaitis E, Bacha F, Nadeau KJ, van Raalte D, Kretzler M, Heerspink H, Bjornstad P. Proteomic Analysis Uncovers Multiprotein Signatures Associated with Early Diabetic Kidney Disease in Youth with Type 2 Diabetes Mellitus. Clin J Am Soc Nephrol. 2024 Dec 1;19(12):1603-1612. doi: 10.2215/CJN.0000000000000559. Epub 2024 Oct 21. PMID 39432369
- [Derived] Lu C, Wolfs D, El Ghormli L, Levitsky LL, Levitt Katz LE, Laffel LM, Patti ME, Isganaitis E. Growth Hormone Mediators and Glycemic Control in Youths With Type 2 Diabetes: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Feb 5;7(2):e240447. doi: 10.1001/jamanetworkopen.2024.0447. PMID 38421647
- [Derived] El Ghormli L, Wen H, Uschner D, Haymond MW, Hughan KS, Kutney K, Laffel L, Tollefsen SE, Escaname EN, Lynch J, Bjornstad P; TODAY Study Group. Trajectories of eGFR and risk of albuminuria in youth with type 2 diabetes: results from the TODAY cohort study. Pediatr Nephrol. 2023 Dec;38(12):4137-4144. doi: 10.1007/s00467-023-06044-3. Epub 2023 Jul 11. PMID 37434027
- [Derived] Levitsky LL, Drews KL, Haymond M, Glubitosi-Klug RA, Levitt Katz LE, Mititelu M, Tamborlane W, Tryggestad JB, Weinstock RS; TODAY Study Group. The obesity paradox: Retinopathy, obesity, and circulating risk markers in youth with type 2 diabetes in the TODAY Study. J Diabetes Complications. 2022 Nov;36(11):108259. doi: 10.1016/j.jdiacomp.2022.108259. Epub 2022 Jul 19. PMID 36150365
- [Derived] Shah AS, Gidding SS, El Ghormli L, Tryggestad JB, Nadeau KJ, Bacha F, Levitt Katz LE, Willi SM, Lima J, Urbina EM; TODAY Study Group. Relationship between Arterial Stiffness and Subsequent Cardiac Structure and Function in Young Adults with Youth-Onset Type 2 Diabetes: Results from the TODAY Study. J Am Soc Echocardiogr. 2022 Jun;35(6):620-628.e4. doi: 10.1016/j.echo.2022.02.001. Epub 2022 Feb 8. PMID 35149207
- [Derived] TODAY Study Group; Shah RD, Braffett BH, Tryggestad JB, Hughan KS, Dhaliwal R, Nadeau KJ, Levitt Katz LE, Gidding SS. Cardiovascular risk factor progression in adolescents and young adults with youth-onset type 2 diabetes. J Diabetes Complications. 2022 Mar;36(3):108123. doi: 10.1016/j.jdiacomp.2021.108123. Epub 2022 Jan 3. PMID 35123868
- [Derived] Trief PM, Uschner D, Tung M, Marcus MD, Rayas M, MacLeish S, Farrell R, Keady J, Chao L, Weinstock RS. Diabetes Distress in Young Adults With Youth-Onset Type 2 Diabetes: TODAY2 Study Results. Diabetes Care. 2022 Mar 1;45(3):529-537. doi: 10.2337/dc21-1689. PMID 35015056
- [Derived] TODAY Study Group; Shah AS, El Ghormli L, Gidding SS, Hughan KS, Levitt Katz LE, Koren D, Tryggestad JB, Bacha F, Braffett BH, Arslanian S, Urbina EM. Longitudinal changes in vascular stiffness and heart rate variability among young adults with youth-onset type 2 diabetes: results from the follow-up observational treatment options for type 2 diabetes in adolescents and youth (TODAY) study. Acta Diabetol. 2022 Feb;59(2):197-205. doi: 10.1007/s00592-021-01796-6. Epub 2021 Sep 20. PMID 34542729
- [Derived] TODAY Study Group. Health Care Coverage and Glycemic Control in Young Adults With Youth-Onset Type 2 Diabetes: Results From the TODAY2 Study. Diabetes Care. 2020 Oct;43(10):2469-2477. doi: 10.2337/dc20-0760. Epub 2020 Aug 10. PMID 32778555
- [Derived] TODAY Study Group. Longitudinal Changes in Cardiac Structure and Function From Adolescence to Young Adulthood in Participants With Type 2 Diabetes Mellitus: The TODAY Follow-Up Study. Circ Heart Fail. 2020 Jun;13(6):e006685. doi: 10.1161/CIRCHEARTFAILURE.119.006685. Epub 2020 Jun 5. PMID 32498621
- [Derived] Saletsky RD, Trief PM, Anderson BJ, Rosenbaum P, Weinstock RS. Parenting style, parent-youth conflict, and medication adherence in youth with type 2 diabetes participating in an intensive lifestyle change intervention. Fam Syst Health. 2014 Jun;32(2):176-85. doi: 10.1037/fsh0000008. Epub 2014 Feb 17. PMID 24548045
- See also: public access to intervention materials used in TODAY — https://today.bsc.gwu.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from July 2004 to February 2009. Participants were recruited from the patient populations of pediatric endocrine clinics at the participating study clinical centers, including satellite clinics. Posters announced the study. Study staff approached youth and their families during medical visits.
Pre-assignment Details: Prior to randomization, eligible subjects entered a 2-6 month run-in period, with goals of weaning from non-study diabetes medications, tolerating metformin at 1000 mg bid but no less than 500 mg bid, attaining glycemic control on metformin alone, mastering standard diabetes education, and adhering to study medication and visit attendance.
Groups:
- 1 Metformin Alone: Metformin alone
  Metformin: capsule, 1000 mg bid, provided encapsulated in weekly packets
- 2 Metformin + Rosliglitazone: Metformin + Rosiglitazone
  Metformin: capsule, 1000 mg bid
  Rosiglitazone: capsule, 4 mg bid, provided encapsulated in weekly packets
- 3 Metformin + Lifestyle Program: Metformin + Lifestyle Program
  Metformin: capsule, 1000 mg bid, encapsulated, provided in weekly packets
  Lifestyle Program: a lifestyle change (LC) phase of weekly sessions for months 1-6, followed by a bi-weekly lifestyle maintenance (LM) phase through months 7-12, and a continued contact (CC) phase from months 13 through the end of the study. The CC phase sessions are scheduled monthly for the initial 12 months (study months 13-24) and then quarterly or 4 times a year to the end of the study
Period: Overall Study
Arm/Group | 1 Metformin Alone | 2 Metformin + Rosliglitazone | 3 Metformin + Lifestyle Program
Started | 232 | 233 | 234
Completed | 232 | 233 | 234
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Age 10-17 years with T2D according to American Diabetes Association criteria for less than 2 years, body mass index (BMI) >=85th percentile, negative diabetes autoantibodies, fasting c-peptide >0.6 ng/mL, and an adult caregiver willing to actively support study participation.
Groups:
- 1 Metformin Alone: Metformin alone
  Metformin: capsule, 1000 mg bid
- 2 Metformin + Rosiglitazone: Metformin + Rosiglitazone
  Metformin: capsule, 1000 mg bid
  Rosiglitazone: capsule, 4 mg bid
- 3 Metformin + Lifestyle Program: Metformin + Lifestyle Program
  Metformin: capsule, 1000 mg bid
  Lifestyle Program: a lifestyle change (LC) phase of weekly sessions for months 1-6, followed by a bi-weekly lifestyle maintenance (LM) phase through months 7-12, and a continued contact (CC) phase from months 13 through the end of the study. The CC phase sessions are scheduled monthly for the initial 12 months (study months 13-24) and then quarterly or 4 times a year to the end of the study
- Total: Total of all reporting groups
Arm/Group | 1 Metformin Alone | 2 Metformin + Rosiglitazone | 3 Metformin + Lifestyle Program | Total
Number analyzed (Participants) | 232 | 233 | 234 | 699
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (1.9) | 14.1 (2.1) | 13.8 (2.0) | 14.0 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 152 | 154 | 452
  Male | 86 | 81 | 80 | 247
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian | 12 | 16 | 13 | 41
  Black Non-Hispanic | 77 | 64 | 86 | 227
  Hispanic | 91 | 101 | 86 | 278
  White Non-Hispanic | 49 | 47 | 46 | 142
  Asian Non-Hispanic | 3 | 5 | 3 | 11
Region of Enrollment [Number; unit: participants]
  United States | 232 | 233 | 234 | 699
Body mass index z-score [Mean (Standard Deviation); unit: z-score] | 2.27 (0.45) | 2.22 (0.49) | 2.18 (0.46) | 2.23 (0.47)
Percent overweight [Mean (Standard Deviation); unit: 100% X (BMI-50th %ile)/50th %ile] | 82.1 (38.3) | 79.1 (38.1) | 75.6 (35.3) | 78.9 (37.3)
Duration of diabetes [Mean (Standard Deviation); unit: months] | 7.8 (6.0) | 8.0 (5.7) | 7.6 (5.8) | 7.8 (5.8)
Total annual household income [Number; unit: participants]
  < $25,000 | 81 | 86 | 92 | 259
  $25,000-49,999 | 83 | 61 | 66 | 210
  >=$50,000 | 44 | 58 | 53 | 155
  unknown | 24 | 28 | 23 | 75
Highest household education level [Number; unit: participants]
  Less than high school | 60 | 60 | 62 | 182
  High school, GED, business or technical | 57 | 49 | 66 | 172
  College no degree | 77 | 78 | 63 | 218
  Graduate degree | 35 | 41 | 38 | 114
  Unknown | 3 | 5 | 5 | 13
Tanner stage by physical examination [Number; unit: participants] — Tanner stage is a standard 5-point scale of pubertal maturity from 1 (pre-pubertal) to 5 (post-pubertal).
  participants
    4 or 5 | 209 | 207 | 204 | 620
    1, 2, or 3 | 23 | 26 | 30 | 79
Nuclear family history of diabetes [Number; unit: participants]
  No | 97 | 93 | 86 | 276
  Yes | 131 | 133 | 143 | 407
  Unknown | 4 | 7 | 5 | 16
Nuclear family + grandparents history of diabetes [Number; unit: participants]
  No | 17 | 26 | 29 | 72
  Yes | 211 | 200 | 200 | 611
  Unknown | 4 | 7 | 5 | 16
Insulin sensitivity (inverse of fasting insulin from OGTT) [Median (Inter-Quartile Range); unit: mL/uU] | .036 [.025 to .050] | .040 [.028 to .064] | .040 [.027 to .067] | .039 [.027 to .060]
Insulinogenic index from OGTT [Median (Inter-Quartile Range); unit: uU/mL divided by mg/dL] | 1.02 [.47 to 1.98] | .92 [.47 to 1.58] | .87 [.47 to 1.89] | .93 [.47 to 1.85]
Body mass index (BMI) [Mean (Standard Deviation); unit: kg per m squared] | 35.8 (8.1) | 35.0 (7.7) | 34.1 (7.1) | 34.9 (7.6)
Waist circumference [Mean (Standard Deviation); unit: cm] | 110.4 (16.6) | 109.0 (17.0) | 106.6 (16.2) | 108.6 (16.7)
Fat mass from DXA [Mean (Standard Deviation); unit: kg] | 33.7 (9.9) | 33.5 (10.2) | 32.6 (9.8) | 33.3 (10.0)
Bone density from DXA [Mean (Standard Deviation); unit: g per cm squared] | 1.09 (.12) | 1.10 (.13) | 1.08 (.12) | 1.09 (.13)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure (Loss of Glycemic Control)
Description: Defined as A1c persistently >=8% over a 6-month period or persistent metabolic decompensation (inability to wean insulin within 3 months of initiation or the occurrence of a second episode within three months of discontinuing insulin)
Time Frame: Study duration - 2 years to 6.5 years of follow up from randomization
Population: The entire cohort of 699 participants was included in the analysis.
Measure: Number; unit: participants
Groups:
- 2 Metformin + Rosliglitazone: Metformin + Rosiglitazone
  Metformin: capsule, 1000 mg bid
  Rosiglitazone: capsule, 4 mg bid
Arm/Group | 1 Metformin Alone | 2 Metformin + Rosliglitazone | 3 Metformin + Lifestyle Program
Number analyzed (Participants) | 232 | 233 | 234
participants
  Treatment failure | 120 | 90 | 109
  Did not fail treatment during trial | 112 | 143 | 125

2. Secondary Outcome: Insulin Sensitivity
Description: All participants were followed to 24 months. Insulin sensitivity is measured from OGTT as inverse of fasting insulin (mL/uU). The analysis sample includes only participants with 24 month data who had not experienced the primary outcome by that time.
Time Frame: 24 months
Population: Participants who were measured at 24 months and had not experienced treatment failure.
Measure: Median (Inter-Quartile Range); unit: mL/uU
Arm/Group | 1 Metformin Alone | 2 Metformin + Rosiglitazone | 3 Metformin + Lifestyle Program
Number analyzed (Participants) | 167 | 157 | 167
mL/uU | 0.037 [0.023 to 0.061] | 0.049 [0.031 to 0.068] | 0.039 [0.027 to 0.064]

3. Secondary Outcome: Number of Serious Adverse Events
Description: Number of serious adverse events reported during the trial. Participant could have multiple episodes reported.
Time Frame: Reported as occurred during study follow-up - 2 years to 6.5 years from randomization.
Population: Entire cohort.
Measure: Number; unit: episodes of serious adverse event
Arm/Group | 1 Metformin Alone | 2 Metformin + Rosiglitazone | 3 Metformin + Lifestyle Program
Number analyzed (Participants) | 232 | 233 | 234
episodes of serious adverse event | 42 | 34 | 58

4. Secondary Outcome: Insulin Secretion
Description: Insulinogenic index determined from OGTT as difference in insulin at 30 minutes minus 0 minutes divided by difference in glucose at 30 minutes minus 0 minutes. The analysis sample includes only participants with 24 month data who had not experienced the primary outcome by that time.
Time Frame: 24 months
Population: Participants who were measured at 24 months and had not experience treatment failure.
Measure: Median (Inter-Quartile Range); unit: uU/mL divided by mg/dL
Arm/Group | 1 Metformin Alone | 2 Metformin + Rosliglitazone | 3 Metformin + Lifestyle Program
Number analyzed (Participants) | 150 | 147 | 155
uU/mL divided by mg/dL | .75 [.33 to 1.39] | .83 [.28 to 1.38] | .71 [.26 to 1.69]

5. Secondary Outcome: Body Composition -- BMI
Description: Body mass index (BMI) measured in kg per meters squared. The analysis sample includes only participants with 24 month data who had not experienced the primary outcome by that time.
Time Frame: 24 months
Population: Cohort measured at 24 months and had not experienced treatment failure.
Measure: Mean (Standard Deviation); unit: kg per meters squared
Arm/Group | 1 Metformin Alone | 2 Metformin + Rosliglitazone | 3 Metformin + Lifestyle Program
Number analyzed (Participants) | 132 | 138 | 134
kg per meters squared | 36.7 (9.1) | 38.2 (8.1) | 35.3 (8.4)

6. Secondary Outcome: Body Composition -- Waist Circumference
Description: Waist circumference (cm) measured at the iliac crest at its outermost point with the measuring tape placed around the participant in a horizontal plane parallel to the floor at the mark and the measurement teken at the end of normal expiration without the tape compressing the skin. The analysis sample includes only participants with 24 month data who had not experienced the primary outcome by that time.
Time Frame: 24 months
Population: Members of cohort measured at 24 months who had not experience treatment failure.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | 1 Metformin Alone | 2 Metformin + Rosliglitazone | 3 Metformin + Lifestyle Program
Number analyzed (Participants) | 132 | 138 | 134
cm | 110.8 (17.5) | 114.0 (16.3) | 108.6 (16.7)

7. Secondary Outcome: Body Composition -- Bone Density
Description: Measured by DXA, both whole body scan and AP-spine scan. The analysis sample includes only participants with 24 month data who had not experienced the primary outcome by that time. In addition, in about 1/3 of participants DXA scans could not be obtained on participants weighing more than 300 pounds (136 kg), the upper limit in size set by the machine manufacturers. Scans were considered invalid if a body part (e.g., arm, leg) was completely off or partially off the scanner, there was hand-hip overlap, or there was motion or movement during the scan.
Time Frame: 24 months
Population: Members of the cohort measured at 24 months who did not experience treatment failure.
Measure: Mean (Standard Deviation); unit: g/cm squared
Arm/Group | 1 Metformin Alone | 2 Metformin + Rosliglitazone | 3 Metformin + Lifestyle Program
Number analyzed (Participants) | 132 | 138 | 134
g/cm squared | 1.15 (.10) | 1.15 (.11) | 1.15 (.12)

8. Secondary Outcome: Body Composition -- Fat Mass
Description: Determined by DXA whole body scan. The analysis sample includes only participants with 24 month data who had not experienced the primary outcome by that time. In addition, in about 1/3 of participants DXA scans could not be obtained on participants weighing more than 300 pounds (136 kg), the upper limit in size set by the machine manufacturers. Scans were considered invalid if a body part (e.g., arm, leg) was completely off or partially off the scanner, there was hand-hip overlap, or there was motion or movement during the scan.
Time Frame: 24 months
Population: Members of the cohort measured at 24 months who did not experience treatment failure.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | 1 Metformin Alone | 2 Metformin + Rosliglitazone | 3 Metformin + Lifestyle Program
Number analyzed (Participants) | 132 | 138 | 134
kg | 36.1 (12.0) | 39.7 (10.5) | 32.2 (9.4)

9. Secondary Outcome: Comorbidity -- Hypertension
Description: A diagnosis was made by an out-of-range value >=95th percentile or systolic >=130 or diastolic >=80 sustained over 6 months or on an anti-hypertensive medication.
Time Frame: Data collected at baseline and during follow-up - 2 years to 6.5 years from randomization.
Population: Entire cohort.
Measure: Number; unit: participants
Arm/Group | 1 Metformin Alone | 2 Metformin + Rosliglitazone | 3 Metformin + Lifestyle Program
Number analyzed (Participants) | 232 | 233 | 234
participants | 57 | 53 | 45

10. Secondary Outcome: Comorbidity -- LDL Dyslipidemia
Description: A diagnosis was made from out-of-range value >= 130 mg/dL sustained over 6 months or put on lipid lowering medication.
Time Frame: Data collected at baseline and during follow-up - 2 years to 6.5 years from randomization.
Population: Entire cohort.
Measure: Number; unit: participants
Arm/Group | 1 Metformin Alone | 2 Metformin + Rosliglitazone | 3 Metformin + Lifestyle Program
Number analyzed (Participants) | 232 | 233 | 234
participants | 18 | 16 | 15

11. Secondary Outcome: Comorbidity -- Triglycerides Dyslipidemia
Description: A diagnosis was made by an out-of-range value >=150 mg/dL sustained over 6 months or on appropriate lipid lowering medication.
Time Frame: Data collected at baseline and during follow-up - 2 years to 6.5 years from randomization.
Population: Entire cohort.
Measure: Number; unit: participants
Arm/Group | 1 Metformin Alone | 2 Metformin + Rosliglitazone | 3 Metformin + Lifestyle Program
Number analyzed (Participants) | 232 | 233 | 234
participants | 20 | 28 | 22

ADVERSE EVENTS:
Time Frame: During the 2-6 month pre-randomization run-in period and during follow-up from 2-6.5 years.
Description: Terminology and criteria standard for clinical trials conducted by NIH were used.
Arm/Group | 1 Metformin Alone | 2 Metformin + Rosliglitazone | 3 Metformin + Lifestyle Program
Serious Adverse Events (participants affected / at risk) | 42/232 | 34/233 | 58/234
Other Adverse Events (participants affected / at risk) | 215/232 | 196/233 | 213/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Metformin Alone (N=232) | 2 Metformin + Rosliglitazone (N=233) | 3 Metformin + Lifestyle Program (N=234)
Diabetic ketoacidosis (Endocrine disorders) | 5 (5) | 3 (3) | 3 (3)
Hyperglycemia (Endocrine disorders) | 3 (3) | 5 (5) | 2 (2)
Hypoglycemia (Endocrine disorders) | 1 (1) | 1 (1) | 2 (2)
Lactic acidosis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
all other (General disorders) | 32 (32) | 25 (25) | 51 (51)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Metformin Alone (N=232) | 2 Metformin + Rosliglitazone (N=233) | 3 Metformin + Lifestyle Program (N=234)
Skin rash on physical examination (Skin and subcutaneous tissue disorders) | 108 (108) | 101 (101) | 95 (95)
Gastrointestinal symptoms (Gastrointestinal disorders) | 129 (129) | 100 (100) | 136 (136) — Frequent stomach pains, bloating, nausea, diarrhea, or loss of appetite.
Edema on physical examination (Skin and subcutaneous tissue disorders) | 17 (17) | 17 (17) | 17 (17)
Hyperglycemia symptoms (Endocrine disorders) | 115 (115) | 98 (98) | 103 (103) — Symptoms of diabetes out of control included nocturia more than once a night on a regular basis, enuresis, increased thirst, urinating more often than usual.
Infection requiring medical attention (Infections and infestations) | 149 (149) | 120 (120) | 151 (151)
Sprain or fracture requiring medical attention (Musculoskeletal and connective tissue disorders) | 66 (66) | 53 (53) | 64 (64)
Muscle ache or pain (Musculoskeletal and connective tissue disorders) | 68 (68) | 53 (53) | 77 (77)
Mild hypoglycemia (Endocrine disorders) | 10 (10) | 19 (19) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This work was conducted by a collaborative group. All investigators in the study group adhere to the Publications & Presentations Policy. The policy spells out procedures for proposing, developing, and submitting publications and presentations using study data. Once results have been published or presented, all members of the study group are free to discuss them.